CLINICAL TRIAL: NCT00979160
Title: Multicenter, Open-Label, Single Arm Phase II Clinical Trial of Dasatinib in the Treatment of Systemic Mastocytosis
Brief Title: Evaluation of Response of Dasatinib to Treat Mastocytosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Prof. Massimo Triggiani, Division of allergy and clinical immunology - University Federico II
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA 180-287
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Patient will be treat at a starting dose of 20mg once daily, that can be escalated up to 100mg once daily.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Starting dosage 20mg once daily, that can be escalated up to 100mg once daily. Patient will remain on treatment for 12 months.
  Other Names: BMS-354825-03

SUMMARY:
This is a multicenter, open-label, single arm phase II non-randomized study of dasatinib in which subjects with systemic mastocytosis (SM) will be treated with a continuous regimen of dasatinib.

Upon completion of a treatment induction period, subjects will be treated with dasatinib at a dose of 100 mg per os (OS) once daily (QD).

DETAILED DESCRIPTION:
Dasatinib may have clinical efficacy and is safe in subjects with SM. This Multicenter, open-label, single arm Phase II study will investigate the clinical response rate in terms of both B/C findings and mediator-related symptoms.

30 adult patients will be treated with a continuous regimen of dasatinib at a starting dose of 20 mg administered orally (PO) once daily (QD), that can be escalated up to 100 mg QD at the end of Week 3. Upon completion of a treatment induction period, subjects will be treated with dasatinib at a daily dose of 100 mg PO QD. Patients will remain on dasatinib treatment for 12 months unless disease progression, unacceptable toxicity or other reasons determine treatment discontinuation. Subjects may continue receiving protocol therapy as long as they are deriving a clinical benefit.

Additionally, all subjects will be followed until disease progression, death, or 12 months beyond discontinuation from study treatment.

The total duration of the study is estimated to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Subjects with confirmed diagnosis of SM according to the WHO criteria and the following must be met:

  * All SM clinical variations, smoldering SM should have ≥ 2 B-findings and severe mediator related symptoms.
  * KIT mutation status on BM cells must be available at baseline or ≤ 6 months prior to study entry.
* Subjects may have not prior treatment with chemotherapeutic regimen including imatinib or have either failed a prior chemotherapeutic regimen including imatinib or other agent.
* At least two weeks must have elapsed from the last dose of chemotherapy, hormonal therapy, immunotherapy, biological therapy or investigational product and radiation therapy, and subjects must have recovered to baseline or Grade ≤ 1 (NCI CTCAE, version 3.0) from the toxicities resulting from any of those recent therapies prior to the first dose of dasatinib.
* ECOG performance status of 0, 1 or 2.
* Subject must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and requirements of the study.
* Adequate liver and renal functions defined as:

  * Total bilirubin ≤ 2 x upper limit of normal (ULN) or ≤ 4 ULN if the sole cause of liver elevation is due to SM
  * AST, ALT and alkaline phosphatase ≤ 2.5 x ULN, or ≤ 5 ULN if the sole cause of liver elevation or bone compromise is due to SM
  * Serum creatinine ≤ 2 x ULN
* Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal.
* Men and women, ages 18 and older.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to at least 4 weeks after the last dose of investigational product.
* Women who are pregnant or breastfeeding
* Indolent SM (presence of B-findings without severe mediator-related symptoms)
* Pericarditis, clinically significant pleural effusion or ascites within 12 months prior to study entry not attributable to SM.
* Pulmonary infiltrates within 4 weeks prior to study entry or abnormal chest X-ray at baseline not attributable to SM.
* Any surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) within 14 days prior to initiation of dasatinib therapy.
* Presence of active bacterial, fungal or viral infections at study entry.
* Clinically significant cardiac disease (NYHA Class III or IV) including preexisting arrhythmia, (such as ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes"), myocardial infarction, uncontrolled angina within 6 months, congestive heart failure, or cardiomyopathy.
* Abnormal QTcF interval prolonged ( ≥ 450 msec) after electrolytes have been corrected on baseline ECG.
* Malabsorption syndrome not attributable to SM or uncontrolled (e.g. not corrected by antimediator therapy) gastrointestinal toxicities (nausea, diarrhea, vomiting) NCI CTCAE Grade = 2.
* Clinically-significant coagulation or platelet function disorder (eg, known von Willebrand's disease).
* Prior or concurrent malignancy, except for the following:

  * Adequately treated basal cell or squamous cell skin cancer.
  * Cervical carcinoma in situ.
  * Adequately treated Stage I or II cancer from which the subject is currently in complete remission.
  * Or any other cancer from which the subject has been disease-free for 3 years.
* Cytopenia(s): ANC <1000/L, or hemoglobin <10 g/dL, or platelets < 100.000/L at study entry unless the pretreatment bone marrow exam and/or presence of disease-related hypersplenism establish that the likely causes of the cytopenia(s) is related to SM.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality, serious uncontrolled medical disorder or active infection that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study.
* Intolerance to dasatinib.
* Administration of hematopoietic growth factors within 14 days prior to study entry.
* Medications that are generally considered to have a risk of causing "Torsades de Pointes"
* Current therapy with steroids must be tapered off within 14 days prior to the start of study medication if it is anticipated that subjects can be tapered off these drugs. Otherwise, for steroid-requiring subjects, investigators should attempt to taper to the minimal dose possible at the time of initiation of dasatinib therapy.
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical response rate in terms of both B/C findings and mediator-related symptoms in subjects with SM who have been treated with dasatinib. | December 2011

SECONDARY OUTCOMES:
To assess of the Time to Response (TTR), Duration of Response (DOR) and Progression-Free survival (PFS). | December 2012
To evaluate the changes in specific biological markers and molecular mutations. | June 2012
To evaluate the safety and toxicity of dasatinib in this population. | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Triggiani, MD, Principal Investigator — Università Federico II
Locations (12):
- Italy (12):
  - Istituto di ematologia "L e A Seragnoli" - Policlinico universitario Sant'Orsola-Malpighi, Bologna
  - Dipartimento di Ematologia - S.O.D. di Ematologia Università degli Studi di Firenze - Azienda Ospedaliera Careggi, Florence
  - Divisione di Ematologia Ospedale Niguarda Ca' Grande, Milan
  - Divisione di Allergologia e Immunologia Clinica, Università Federico II, Napoli
  - Divisione di Ematologia Università di Torino Ospedale San Luigi Gonzaga, Orbassano (TO)
  - Istituto di Ematologia Università degli Studi di Pavia - Policlinico S. Matteo IRCCS, Pavia
  - Unità di Ematologia e Trapianto Osseo CROB, Centro di Riferimento Oncologico di Basilicata +39 0972 726729 Fax +30 0972 726217 e-mail: p.musto@crob.it, Rionero in Vulture (Pz)
  - Ematologia Tor Vergata University Hospital, Roma
  - Divisione di Ematologia Policlinico Universitario "Agostino Gemelli", Roma
  - Ematologia e Trapianti Università degli Studi di Siena - Policlinico S. Maria alle Scotte, Siena
  - Divisione di Ematologia e Trapianto Midollo Osseo Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine
  - Sezione di Ematologia - Dipartimento di Medicina Clinica e Sperimentale Policlinico G.B.Rossi - Università degli Studi di Verona, Verona